CLINICAL TRIAL: NCT05425732
Title: A Phase 3, Randomized, Double-blind, Active Comparator-controlled Clinical Study to Evaluate the Safety, Tolerability, and Immunogenicity of V116 in Pneumococcal Vaccine-naïve Adults
Brief Title: Safety and Immunogenicity of V116 in Pneumococcal Vaccine-naïve Adults (V116-003, STRIDE-3)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V116-003; V116-003 (Other: MSD); 2022-000258-27 (EudraCT Number)
Record Dates: First submitted 2022-06-15; First posted 2022-06-21 (Actual); Results first posted 2024-06-10 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Pneumococcal Infection
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 V116 (Experimental): Pneumococcal vaccine-naïve adult participants (≥50 years of age) receive a single dose of V116 on Day 1.
  Interventions: Biological: V116
- Cohort 1 PCV20 (Active Comparator): Pneumococcal vaccine-naïve adult participants (≥50 years of age) receive a single dose of PCV20 on Day 1.
  Interventions: Biological: PCV20
- Cohort 2 V116 (Experimental): Pneumococcal vaccine-naïve adult participants (18 to 49 years of age) receive a single dose of V116 on Day 1.
  Interventions: Biological: V116
- Cohort 2 PCV20 (Active Comparator): Pneumococcal vaccine-naïve adult participants (18 to 49 years of age) receive a single dose of PCV20 on Day 1.
  Interventions: Biological: PCV20

INTERVENTIONS:
Biological: V116 — 0.5 mL injection solution in prefilled syringe containing 4 μg of each PnPs antigen (3, 6A, 7F, 8, 9N, 10A, 11A, 12F, 15A, 15C, 16F, 17F, 19A, 20A, 22F, 23A, 23B, 24F, 31, 33F, and 35B) given by intramuscular (IM) injection.
  Other Names: Pneumococcal 21-valent Conjugate Vaccine
  Arms: Cohort 1 V116; Cohort 2 V116
Biological: PCV20 — 0.5 mL injection suspension in prefilled syringe containing 2.2 μg of each PnPs antigen (1, 3, 4, 5, 6A, 7F, 8, 9V, 10A, 11A, 12F, 14, 15B, 18C, 19A, 19F, 22F, 23F, 33F) and 4.4 μg of PnPs antigen 6B.
  Other Names: Prevnar 20™; APEXXNAR™
  Arms: Cohort 1 PCV20; Cohort 2 PCV20

SUMMARY:
This is a phase 3, randomized, double-blind, active comparator-controlled study of the safety, tolerability, and immunogenicity of V116 compared to PCV20 (pneumococcal 20-valent conjugate vaccine ([Prevnar 20™ / APEXXNAR™]) in pneumococcal vaccine-naïve adults. It is hypothesized that V116 is noninferior to PCV20 for the common serotypes and superior to PCV20 for the unique serotypes as assessed by serotype specific opsonophagocytic activity (OPA) 30 days postvaccination. It is also hypothesized that V116 in participants 18 to 49 years of age immunobridges to V116 in participants 50 to 64 years of age as assessed by serotype specific OPA geometric mean titers (GMTs) 30 days postvaccination for all 21 serotypes in V116. Participants ≥50 years of age will be enrolled in Cohort 1, and participants 18 to 49 years of age will be enrolled in Cohort 2.

ELIGIBILITY:
Inclusion Criteria:

* For females, is not pregnant or breastfeeding and is either not a woman of childbearing potential (WOCBP) or is a WOCBP and uses acceptable contraception/abstinence; and has medical, menstrual, and recent sexual activity history reviewed by the investigator to decrease the chance of an early undetected pregnancy.

Exclusion Criteria:

* Has a history of invasive pneumococcal disease (IPD) [positive blood culture, positive cerebrospinal fluid culture, or positive culture at another sterile site] or known history of other culture-positive pneumococcal disease within 3 years of Visit 1 (Day 1)
* Has a known hypersensitivity to any component of V116 or PCV20, including diphtheria toxoid
* Has a known or suspected impairment of immunological function including, but not limited to, a history of congenital or acquired immunodeficiency, documented human immunodeficiency virus (HIV) infection, functional or anatomic asplenia, or history of autoimmune disease
* Has a coagulation disorder contraindicating IM vaccination
* Had a recent febrile illness (defined as oral or tympanic temperature ≥100.4°F [≥38.0°C] or axillary or temporal temperature ≥99.4°F [≥37.4°C]) or received antibiotic therapy for any acute illness occurring <72 hours before receipt of study vaccine
* Has a known malignancy that is progressing or has required active treatment <3 years before enrollment
* Received prior administration (prior to age of 5 is acceptable) of any pneumococcal vaccine or is expected to receive any pneumococcal vaccine during the study outside the protocol
* Received systemic corticosteroids (prednisone equivalent of ≥20 mg/day) for ≥14 consecutive days and has not completed intervention ≥14 days before receipt of study vaccine
* Is currently receiving immunosuppressive therapy, including chemotherapeutic agents or other immunotherapies/immunomodulators used to treat cancer or other conditions, and interventions associated with organ or bone marrow transplantation, or autoimmune disease
* Received any nonlive vaccine ≤14 days before receipt of study vaccine or is scheduled to receive any nonlive vaccine ≤30 days after receipt of study vaccine (inactivated influenza and SARS-CoV2 vaccines may be acceptable)
* Received any live virus vaccine ≤30 days before receipt of study vaccine or is scheduled to receive any live virus vaccine ≤30 days after receipt of study vaccine
* Received a blood transfusion or blood products, including immunoglobulin ≤6 months before receipt of study vaccine or is scheduled to receive a blood transfusion or blood product until the Day 30 postvaccination blood draw is complete

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2663 (Actual)
Dates: Start 2022-07-13 (Actual); Primary Completion 2023-05-18 (Actual); Study Completion 2023-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (112):
- United States (60):
  - Central Research Associates ( Site 0067), Birmingham, Alabama
  - Lenzmeier Family Medicine/CCT Research ( Site 0006), Glendale, Arizona
  - Desert Clinical Research/ CCT Research ( Site 0040), Mesa, Arizona
  - Foothills Research Center/ CCT Research ( Site 0021), Phoenix, Arizona
  - Fiel Family and Sports Medicine, PC/CCT Research ( Site 0003), Tempe, Arizona
  - Baptist Health Center For Clinical Research ( Site 0019), Little Rock, Arkansas
  - Southland Clinical Research Center-Research ( Site 0054), Fountain Valley, California
  - Sunwise Clinical Research ( Site 0024), Lafayette, California
  - Chemidox Clinical Trials ( Site 0048), Lancaster, California
  - Paradigm Clinical Research Centers, Inc ( Site 0018), Redding, California
  - Peninsula Research Associates ( Site 0079), Rolling Hills Estates, California
  - Acclaim Clinical Research ( Site 0083), San Diego, California
  - Millennium Clinical Trials ( Site 0013), Simi Valley, California
  - Lynn Institute of Denver ( Site 0012), Aurora, Colorado
  - Paradigm Clinical Research Centers, Inc ( Site 0027), Wheat Ridge, Colorado
  - JEM Research Institute ( Site 0072), Atlantis, Florida
  - Alliance for Multispecialty Research, LLC ( Site 0015), Coral Gables, Florida
  - Hillcrest Medical Research ( Site 0049), DeLand, Florida
  - East Coast Institute for Research, LLC ( Site 0070), Jacksonville, Florida
  - East Coast Institute for Research ( Site 0071), Lake City, Florida
  - L&C Professional Medical Research Institute ( Site 0025), Miami, Florida
  - Advanced Medical Research Institute ( Site 0014), Miami, Florida
  - Headlands Research Orlando ( Site 0031), Orlando, Florida
  - Genesis Clinical Research, LLC ( Site 0016), Tampa, Florida
  - Clinical Research Trials of Florida ( Site 0007), Tampa, Florida
  - Palm Beach Research Center ( Site 0060), West Palm Beach, Florida
  - Clinical Research Prime ( Site 0010), Idaho Falls, Idaho
  - Solaris Clinical Research ( Site 0008), Meridian, Idaho
  - Versailles Family Medicine / CCT Research ( Site 0063), Versailles, Kentucky
  - Arcturus Healthcare , PLC, Troy Internal Medicine Research Division ( Site 0038), Troy, Michigan
  - Alliance for Multispecialty Research, LLC ( Site 0026), Kansas City, Missouri
  - Skyline Medical Center/CCT Research ( Site 0028), Elkhorn, Nebraska
  - Methodist Physicians Clinic/CCT Research ( Site 0058), Fremont, Nebraska
  - Meridian Clinical Research, LLC ( Site 0045), Norfolk, Nebraska
  - Healor Primary Care / CCT Research ( Site 0056), Las Vegas, Nevada
  - Excel Clinical Research, LLC ( Site 0077), Las Vegas, Nevada
  - Santa Rosa Medical Centers of Nevada / CCT Research ( Site 0029), Las Vegas, Nevada
  - Smith Allergy & Asthma Specialists-Corning Center for Clinical Research ( Site 0032), Horseheads, New York
  - Aventiv Research Inc ( Site 0044), Columbus, Ohio
  - Advanced Medical Research ( Site 0002), Maumee, Ohio
  - Lynn Institute of Norman ( Site 0001), Norman, Oklahoma
  - Lynn Health Science Institute ( Site 0005), Oklahoma City, Oklahoma
  - Lynn Institute of Tulsa ( Site 0084), Tulsa, Oklahoma
  - Summit Headlands ( Site 0047), Portland, Oregon
  - Velocity Clinical Research, Greenville ( Site 0043), Greenville, South Carolina
  - Trial Management Associates ( Site 0089), Myrtle Beach, South Carolina
  - Tekton Research, Inc. ( Site 0053), Austin, Texas
  - WR-Global Medical Research, LLC ( Site 0065), Dallas, Texas
  - Elixir Research Group - W Houston ( Site 0068), Houston, Texas
  - Epic Clinical Research ( Site 0082), Lewisville, Texas
  - DCOL Center for Clinical Research ( Site 0051), Longview, Texas
  - Research Your Health ( Site 0042), Plano, Texas
  - IMA Clinical Research San Antonio ( Site 0009), San Antonio, Texas
  - VIP Trials ( Site 0086), San Antonio, Texas
  - Dynamed Clinical Research, LP d/b/a DM Clinical Research-DM Clinical Research ( Site 0036), Tomball, Texas
  - Olympus Family Medicine/CCT Research ( Site 0074), Holladay, Utah
  - South Ogden Family Medicine/ CCT Research ( Site 0022), Ogden, Utah
  - Charlottesville Medical Research ( Site 0034), Charlottesville, Virginia
  - Health Research of Hampton Roads, Inc. ( Site 0004), Newport News, Virginia
  - MultiCare Rockwood Cheney Clinic ( Site 0037), Spokane, Washington
- Australia (5):
  - Paratus Clinical Research Canberra ( Site 3000), Bruce, Australian Capital Territory
  - Emeritus Research ( Site 3004), Botany, New South Wales
  - Paratus Clinical Research Central Coast ( Site 3001), Kanwal, New South Wales
  - Westmead Hospital ( Site 3005), Westmead, New South Wales
  - Emeritus Research ( Site 3003), Camberwell, Victoria
- Belgium (2):
  - Anima Diepenbeek ( Site 1003), Diepenbeek, Limburg
  - Private Practice - Dr. Martinot Jean-Benoit ( Site 1001), Erpent, Namur
- Chile (4):
  - Universidad San Sebastian - Providencia ( Site 0514), Providencia, Region M. de Santiago
  - Espacio Eme ( Site 0509), Santiago, Region M. de Santiago
  - Centro de Investigacion Clinicadela Universidad Catolica ( Site 0503), Santiago, Region M. de Santiago
  - Hospital hernan henriquez aravena de temuco-Unidad de Investigación Clínica ( Site 0504), Temuco, Región de la Araucanía
- Germany (6):
  - InfektioResearch ( Site 1203), Frankfurt am Main, Hesse
  - Universitaetsklinikum Koeln ( Site 1206), Cologne, North Rhine-Westphalia
  - Medizentrum Essen Borbeck ( Site 1200), Essen, North Rhine-Westphalia
  - Novopraxis Berlin GbR ( Site 1201), Berlin
  - Universitaetsklinikum Hamburg-Eppendorf-Infektiologie ( Site 1202), Hamburg
  - Hamburger Institut fuer Therapieforschung GmbH ( Site 1204), Hamburg
- New Zealand (5):
  - Lakeland Clinical Trials ( Site 3102), Rotorua, Bay of Plenty
  - P3 Research - Tauranga ( Site 3100), Tauranga, Bay of Plenty
  - Southern Clinical Trials Ltd ( Site 3104), Christchurch, Canterbury
  - Southern Clinical Trials Waitemata Ltd ( Site 3105), Auckland
  - P3 Research - Wellington ( Site 3101), Wellington
- Puerto Rico (5):
  - Cooperativa De Facultad Medica Sanacoop-Instituto Sanacoop ( Site 0601), Bayamón
  - San Juan Bautista School of Medicine - Clinical Research Unit ( Site 0606), Caguas
  - Clinical Research Investigator Group ( Site 0611), Canovanas
  - Ponce School Of Medicine Caimed Center ( Site 0602), Ponce
  - Clinical Research Puerto Rico ( Site 0600), San Juan
- South Korea (12):
  - Gachon University Gil Medical Center ( Site 3205), Namdong-gu, Incheon
  - Korea University Ansan Hospital ( Site 3201), Ansan-si, Kyonggi-do
  - The Catholic University Of Korea St. Vincent's Hospital-Internal Medicine ( Site 3206), Suwon, Kyonggi-do
  - Ajou University Hospital-Department of Infectious Diseases ( Site 3209), Suwon, Kyonggi-do
  - Kyungpook National University Chilgok Hospital-Division of Infectious Diseases ( Site 3207), Deagu, Taegu-Kwangyokshi
  - The Catholic University of Korea, Eunpyeong St. Mary's Hospital ( Site 3202), Seoul
  - Severance Hospital, Yonsei University Health System-Division of Infectious Diseases ( Site 3210), Seoul
  - Samsung Medical Center ( Site 3211), Seoul
  - The Catholic Univ. of Korea Seoul St. Mary's Hospital ( Site 3203), Seoul
  - Hallym University Kangnam Sacred Heart Hospital-Internal Medicine ( Site 3204), Seoul
  - Ewha Womans University Mokdong Hospital-Infectious Diseases ( Site 3208), Seoul
  - Korea University Guro Hospital ( Site 3200), Seoul
- Sweden (5):
  - ProbarE ( Site 1400), Lund, Skåne County
  - CTC Karolinska ( Site 1405), Solna, Stockholm County
  - ProbarE i Stockholm AB ( Site 1401), Stockholm, Stockholm County
  - Studieenheten Akademiskt Specialistcentrum ( Site 1403), Stockholm, Stockholm County
  - CTC MTC ( Site 1404), Uppsala, Uppsala County
- Taiwan (4):
  - National Cheng Kung University Hospital ( Site 3301), Tainan
  - National Taiwan University Hospital ( Site 3300), Taipei
  - Taipei Medical University Hospital ( Site 3302), Taipei
  - Chang Gung Medical Foundation-Linkou Branch ( Site 3303), Taoyuan District
- Turkey (Türkiye) (4):
  - Sakarya Training and Research Hospital ( Site 2205), Adapazarı, Sakarya
  - Hacettepe Universite Hastaneleri ( Site 2204), Ankara
  - Ankara City Hospital ( Site 2200), Ankara
  - Acibadem Universitesi Atakent Hastanesi-Infectious Disease ( Site 2201), Istanbul

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Platt HL, Bruno C, Buntinx E, Pelayo E, Garcia-Huidobro D, Barranco-Santana EA, Sjoberg F, Song JY, Grijalva CG, Orenstein WA, Morgan L, Fernsler D, Xu W, Waleed M, Li J, Buchwald UK; STRIDE-3 Study Group. Safety, tolerability, and immunogenicity of an adult pneumococcal conjugate vaccine, V116 (STRIDE-3): a randomised, double-blind, active comparator controlled, international phase 3 trial. Lancet Infect Dis. 2024 Oct;24(10):1141-1150. doi: 10.1016/S1473-3099(24)00344-X. Epub 2024 Jul 1. PMID 38964361
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26092&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Pneumococcal vaccine-naïve adults ≥18 years of age were enrolled in this study. Participants with underlying chronic conditions were eligible if the conditions were assessed to be stable per the investigator's judgment.
Groups:
- Cohort 1 V116: Pneumococcal vaccine-naïve adult participants (≥50 years of age) receive a single dose of pneumococcal 21-valent conjugate vaccine (V116) on Day 1.
- Cohort 1 PCV20: Pneumococcal vaccine-naïve adult participants (≥50 years of age) receive a single dose of pneumococcal 20-valent conjugate vaccine (PCV20) on Day 1.
Period: Overall Study
Arm/Group | Cohort 1 V116 | Cohort 1 PCV20 | Cohort 2 V116 | Cohort 2 PCV20
Started (Randomized participants) | 1181 (Includes two participants with unplanned randomization to both PCV20 and V116) | 1181 (Includes two participants with unplanned randomization to both PCV20 and V116) | 201 | 100
Vaccinated (Randomized participants who were vaccinated) | 1179 (Includes two participants with unplanned vaccination with both PCV20 and V116) | 1177 (Includes two participants with unplanned vaccination with both PCV20 and V116) | 200 | 100
Safety All Cause Mortality (ACM) Population | 1179 (.The two participants with unplanned randomization and vaccination with both V116 and PCV20 are excluded from the ACM population) | 1179 (The two participants with unplanned randomization and vaccination with both V116 and PCV20 are excluded from the ACM population) | 201 | 100
All Participants As Treated (APaT) (Randomized participants who were included in the group corresponding to the vaccine they actually received) | 1177 (The two participants with unplanned randomization to both the V116 and PCV20 treatment groups were excluded from the All Participants As Treated population.) | 1175 (The two participants with unplanned randomization to both the V116 and PCV20 treatment groups were excluded from the All Participant As Treated population.) | 200 | 100
Safety Adverse Event (AE) Population (All Participants As Treated (APaT)) | 1177 | 1175 | 200 | 100
Completed | 1160 | 1152 | 195 | 96
Not Completed | 21 | 29 | 6 | 4
Not completed — Death | 4 | 2 | 0 | 0
Not completed — Lost to Follow-up | 10 | 15 | 5 | 3
Not completed — Physician Decision | 0 | 2 | 0 | 0
Not completed — Randomized By Mistake Without Study Treatment | 1 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 8 | 1 | 1
Not completed — Randomized to PCV20 first, discontinued; then randomized to V116 second | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All vaccinated participants. Includes two participants from Cohort 1 who had unplanned vaccinations with both V116 and PCV20
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 V116 | Cohort 1 PCV20 | Cohort 2 V116 | Cohort 2 PCV20 | Total
Number analyzed (Participants) | 1179 | 1177 | 200 | 100 | 2656
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.9 (8.3) | 63.9 (8.3) | 35.2 (9.0) | 34.6 (8.7) | 60.7 (12.4)
Age, Customized [Number; unit: Participants]
  18 to 49 years | 0 | 0 | 200 | 100 | 300
  50 to 64 years | 589 | 587 | 0 | 0 | 1176
  65 to 74 years | 464 | 464 | 0 | 0 | 928
  75 to 84 years | 112 | 113 | 0 | 0 | 225
  ≥85 years | 14 | 13 | 0 | 0 | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 687 | 670 | 137 | 64 | 1558
  Male | 492 | 507 | 63 | 36 | 1098
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 259 | 242 | 58 | 24 | 583
  Not Hispanic or Latino | 909 | 922 | 141 | 76 | 2048
  Unknown or Not Reported | 11 | 13 | 1 | 0 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 4 | 0 | 1 | 9
  Asian | 148 | 168 | 38 | 15 | 369
  Native Hawaiian or Other Pacific Islander | 17 | 16 | 1 | 2 | 36
  Black or African American | 116 | 115 | 13 | 14 | 258
  White | 867 | 844 | 139 | 62 | 1912
  More than one race | 26 | 30 | 9 | 6 | 71
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Solicited Injection-site Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Solicited injection-site AEs consist of the following: pain/tenderness, redness/erythema, and swelling.
Time Frame: Up to 5 days post-vaccination
Population: All participants as treated consisting of randomized participants who were included in the group corresponding to the vaccine actually received.
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1 V116 | Cohort 1 PCV20 | Cohort 2 V116 | Cohort 2 PCV20
Number analyzed (Participants) | 1177 | 1175 | 200 | 100
Percentage of participants
  Injection site erythema | 5.4 | 6.3 | 15.5 | 13.0
  Injection site pain | 39.4 | 51.7 | 71.5 | 74.0
  Injection site swelling | 6.0 | 8.3 | 14.0 | 14.0
Statistical Analysis 1: Comparison: Cohort 1 V116 vs Cohort 1 PCV20; Injection site erythema: estimated difference in percent; Test type: Other — Miettinen & Nurminen method; Difference in Percent = -0.9, 96% CI 2-sided [-2.8 to 1.1] — V116 minus PCV20
Statistical Analysis 2: Comparison: Cohort 1 V116 vs Cohort 1 PCV20; Injection site pain: estimated difference in percent; Test type: Other — Miettinen & Nurminen method; Difference in Percent = -12.2, 95% CI 2-sided [-16.2 to -8.2] — V116 minus PCV20
Statistical Analysis 3: Comparison: Cohort 1 V116 vs Cohort 1 PCV20; Injection site swelling: estimated difference in percent; Test type: Other — Miettinen & Nurminen method; Difference in Percent = -2.3, 95% CI 2-sided [-4.4 to -0.2] — V116 minus PCV20
Statistical Analysis 4: Comparison: Cohort 2 V116 vs Cohort 2 PCV20; Injection site erythema: estimated difference in percent; Test type: Other — Miettinen & Nurminen method; Difference in Percent = 2.5, 95% CI 2-sided [-6.6 to 10.3] — V116 minus PCV20
Statistical Analysis 5: Comparison: Cohort 2 V116 vs Cohort 2 PCV20; Injection site pain: estimated difference in percent; Test type: Other — Miettinen & Nurminen method; Difference in Percent = -2.5, 95% CI 2-sided [-12.7 to 8.6] — V116 minus PCV20
Statistical Analysis 6: Comparison: Cohort 2 V116 vs Cohort 2 PCV20; Injection site swelling: estimated difference in percent; Test type: Other — Miettinen & Nurminen method; Difference in Percent = 0.0, 95% CI 2-sided [-9.2 to 7.9] — V116 minus PCV20

2. Primary Outcome: Percentage of Participants With Solicited Systemic AEs
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Solicited systemic AEs consist of the following: fatigue (tiredness), headache, myalgia (muscle aches), and pyrexia (maximum temperature ≥ 100.4 °F/38.0 °C)
Time Frame: Up to 5 days post-vaccination
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1 V116 | Cohort 1 PCV20 | Cohort 2 V116 | Cohort 2 PCV20
Number analyzed (Participants) | 1177 | 1175 | 200 | 100
Percentage of participants
  Fatigue | 20.1 | 19.6 | 40.5 | 34.0
  Headache | 11.5 | 12.9 | 29.5 | 24.0
  Myalgia | 5.9 | 6.7 | 16.5 | 14.0
  Pyrexia | 1.3 | 1.3 | 3.5 | 1.0
Statistical Analysis 1: Comparison: Cohort 1 V116 vs Cohort 1 PCV20; Fatigue: estimated difference in percent; Test type: Other — Miettinen & Nurminen method; Difference in Percent = 0.6, 95% CI 2-sided [-2.7 to 3.8] — V116 minus PCV20
Statistical Analysis 2: Comparison: Cohort 1 V116 vs Cohort 1 PCV20; Headache: estimated difference in percent; Test type: Other — Miettinen & Nurminen method; Difference in Percent = -1.5, 95% CI 2-sided [-4.1 to 1.2] — V116 minus PCV20
Statistical Analysis 3: Comparison: Cohort 1 V116 vs Cohort 1 PCV20; Myalgia: estimated difference in percent; Test type: Other — Miettinen & Nurminen method; Difference in Percent = -0.8, 96% CI 2-sided [-2.8 to 1.2] — V116 minus PCV20
Statistical Analysis 4: Comparison: Cohort 1 V116 vs Cohort 1 PCV20; Pyrexia: estimated difference in percent; Test type: Other — Miettinen & Nurminen method; Difference in Percent = -0.0, 95% CI 2-sided [-1.0 to 1.0] — V116 minus PCV20
Statistical Analysis 5: Comparison: Cohort 2 V116 vs Cohort 2 PCV20; Fatigue: estimated difference in percent; Test type: Other — Miettinen & Nurminen method; Difference in Percent = 6.5, 95% CI 2-sided [-5.3 to 17.6] — V116 minus PCV20
Statistical Analysis 6: Comparison: Cohort 2 V116 vs Cohort 2 PCV20; Headache: estimated difference in percent; Test type: Other — Miettinen & Nurminen method; Difference in Percent = 5.5, 05% CI 2-sided [-5.5 to 15.5] — V116 minus PCV20
Statistical Analysis 7: Comparison: Cohort 2 V116 vs Cohort 2 PCV20; Myalgia: estimated difference in percent; Test type: Other — Miettinen & Nurminen method; Difference in Percent = 2.5, 95% CI 2-sided [-6.8 to 10.6] — V116 minus PCV20
Statistical Analysis 8: Comparison: Cohort 2 V116 vs Cohort 2 PCV20; Pyrexia: estimated difference in percent; Test type: Other — Miettinen & Nurminen method; Difference in Percent = 2.5, 95% CI 2-sided [-2.2 to 6.2] — V116 minus PCV20

3. Primary Outcome: Percentage of Participants With Vaccine-related Serious AE (SAE)
Description: A vaccine-related SAE is any untoward medical consequence that results in death, is life-threatening, requires inpatient hospitalization or prolongs existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is an other important medical event, which is determined by the investigator to be related to the vaccine.
Time Frame: Up to 194 days post-vaccination
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1 V116 | Cohort 1 PCV20 | Cohort 2 V116 | Cohort 2 PCV20
Number analyzed (Participants) | 1177 | 1175 | 200 | 100
Percentage of participants | 0.0 | 0.0 | 0.0 | 0.0

4. Primary Outcome: Serotype Specific Opsonophagocytic (OPA) Geometric Mean Titers (GMTs) in Cohort 1 Only, for the Pneumococcal Serotypes Contained in V116 and PCV20
Description: The serotype specific OPA GMTs for the pneumococcal serotypes in cohort 1 of V116 and PCV20 only were determined using the multiplex opsonophagocytic assay (MOPA). GMT values were estimated from a constrained longitudinal data analysis; (cLDA) model. Per protocol, within group, confidence intervals (CIs) or any other measures of dispersion were not planned or determined. The 10 common pneumococcal serotypes in both V116 and PCV20 were as follows: 3, 6A, 7F, 8, 10A, 11A, 12F, 19A, 22F, and 33F. The 11 unique pneumococcal serotypes in V116 were as follows: 9N, 15A, 15C, 16F, 17F, 20A, 23A, 23B, 24F, 31, and 35B. Per protocol, Cohort 2 were not analyzed in this outcome measure.
Time Frame: Day 30 post-vaccination
Population: All randomized participants from cohort 1 only, without deviations from the protocol that may substantially affect immunogenicity. Deviations include, but are not limited to the following: missing serology results; and blood draw out of window. Per protocol, Cohort 2 were not analyzed in this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Cohort 1 V116 | Cohort 1 PCV20 | Cohort 2 V116 | Cohort 2 PCV20
Number analyzed (Participants) | 1179 | 1177 | 0 | 0
Titer
  Serotype 3: number analyzed (Participants) | 1154 | 1161 | 0 | 0
  Serotype 3 | 274.0 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 176.7 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 6A: number analyzed (Participants) | 1148 | 1153 | 0 | 0
  Serotype 6A | 2302.0 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 2972.5 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 7F: number analyzed (Participants) | 1152 | 1158 | 0 | 0
  Serotype 7F | 3637.4 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 3429.9 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 8: number analyzed (Participants) | 1155 | 1158 | 0 | 0
  Serotype 8 | 2501.3 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 1811.1 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 10A: number analyzed (Participants) | 1161 | 1159 | 0 | 0
  Serotype 10A | 3893.4 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 4678.0 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 11A: number analyzed (Participants) | 1145 | 1150 | 0 | 0
  Serotype 11A | 3232.6 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 2092.8 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 12F: number analyzed (Participants) | 1160 | 1161 | 0 | 0
  Serotype 12F | 2641.2 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 2499.6 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 19A: number analyzed (Participants) | 1159 | 1162 | 0 | 0
  Serotype 19A | 2136.1 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 2817.8 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 22F: number analyzed (Participants) | 1147 | 1154 | 0 | 0
  Serotype 22F | 3874.5 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 4770.1 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 33F: number analyzed (Participants) | 1154 | 1157 | 0 | 0
  Serotype 33F | 13558.9 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 11742.1 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 9N: number analyzed (Participants) | 1147 | 1150 | 0 | 0
  Serotype 9N | 7470.7 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 1640.4 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype15A: number analyzed (Participants) | 1107 | 1102 | 0 | 0
  Serotype15A | 5237.2 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 1589.0 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 15C: number analyzed (Participants) | 1153 | 1158 | 0 | 0
  Serotype 15C | 4216.2 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 2072.3 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 16F: number analyzed (Participants) | 1151 | 1153 | 0 | 0
  Serotype 16F | 4868.2 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 846.3 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined.. |  |
  Serotype 17F: number analyzed (Participants) | 1148 | 1156 | 0 | 0
  Serotype 17F | 7764.9 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 460.4 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 20A: number analyzed (Participants) | 1161 | 1155 | 0 | 0
  Serotype 20A | 6099.2 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 631.1 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 23A: number analyzed (Participants) | 1132 | 1104 | 0 | 0
  Serotype 23A | 3737.2 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 461.5 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 23B: number analyzed (Participants) | 1160 | 1160 | 0 | 0
  Serotype 23B | 1082.5 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 107.3 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 24F: number analyzed (Participants) | 1153 | 1130 | 0 | 0
  Serotype 24F | 2728.6 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 70.5 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 31: number analyzed (Participants) | 1153 | 1154 | 0 | 0
  Serotype 31 | 3132.5 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 144.4 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 35B: number analyzed (Participants) | 1153 | 1159 | 0 | 0
  Serotype 35B | 8527.8 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 1383.0 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
Statistical Analysis 1: Comparison: Cohort 1 V116 vs Cohort 1 PCV20; Serotype 3: V116/PCV20 GMT Ratio; Test type: Non-Inferiority — A conclusion of non-inferiority is based on the lower bound of the 95% CI for the estimated GMT Ratio (V116/PCV20) being > 0.5 (one-sided p-value < 0.025); p < 0.001, cLDA model — 1-sided; GMT Ratio = 1.55, 95% CI 2-sided [1.40 to 1.72] — V116/PCV20
Statistical Analysis 2: Comparison: Cohort 1 V116 vs Cohort 1 PCV20; Serotype 6A: V116/PCV20 GMT Ratio; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, cLDA model; GMT Ratio = 0.77, 95% CI 2-sided [0.68 to 0.88] — V116/PCV20
Statistical Analysis 3: Comparison: Cohort 1 V116 vs Cohort 1 PCV20; Serotype 7F: V116/PCV20 GMT Ratio; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, cLDA model; GMT Ratio = 1.06, 95% CI 2-sided [0.95 to 1.18] — V116/PCV20
Statistical Analysis 4: Comparison: Cohort 1 V116 vs Cohort 1 PCV20; Serotype 8: V116/PCV20 GMT Ratio; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, cLDA model; GMT Ratio = 1.38, 95% CI 2-sided [1.25 to 1.53] — V116/PCV20
Statistical Analysis 5: Comparison: Cohort 1 V116 vs Cohort 1 PCV20; Serotype 10A: V116/PCV20 GMT Ratio; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, cLDA model; GMT Ratio = 0.83, 95% CI 2-sided [0.75 to 0.93] — V116/PCV20
Statistical Analysis 6: Comparison: Cohort 1 V116 vs Cohort 1 PCV20; Serotype 11A: V116/PCV20 GMT Ratio; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, cLDA model; GMT Ratio = 1.54, 95% CI 2-sided [1.39 to 1.72] — V116/PCV20
Statistical Analysis 7: Comparison: Cohort 1 V116 vs Cohort 1 PCV20; Serotype 12F: V116/PCV20 GMT Ratio; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, cLDA model; GMT Ratio = 1.06, 95% CI 2-sided [0.92 to 1.21] — V116/PCV20
Statistical Analysis 8: Comparison: Cohort 1 V116 vs Cohort 1 PCV20; Serotype 19A: V116/PCV20 GMT Ratio; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, cLDA model; GMT Ratio = 0.76, 95% CI 2-sided [0.69 to 0.84] — V116/PCV20
Statistical Analysis 9: Comparison: Cohort 1 V116 vs Cohort 1 PCV20; Serotype 22F: V116/PCV20 GMT Ratio; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, cLDA model; GMT Ratio = 0.81, 95% CI 2-sided [0.72 to 0.92] — V116/PCV20
Statistical Analysis 10: Comparison: Cohort 1 V116 vs Cohort 1 PCV20; Serotype 33F: V116/PCV20 GMT Ratio; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, cLDA model; GMT Ratio = 1.15, 95% CI 2-sided [1.01 to 1.32] — V116/PCV20
Statistical Analysis 11: Comparison: Cohort 1 V116 vs Cohort 1 PCV20; Serotype 9N: V116/PCV20 GMT Ratio; Test type: Superiority — A conclusion of superiority is based on the lower bound of the 95% CI for the estimated GMT ratio (V116/PCV20) being > 2.0 (one-sided p-value < 0.025); p < 0.001, cLDA model; GMT Ratio = 4.55, 95% CI 2-sided [4.12 to 5.04] — V116/PCV20
Statistical Analysis 12: Comparison: Cohort 1 V116 vs Cohort 1 PCV20; Serotype 15A: V116/PCV20 GMT Ratio; Test type: Superiority — [test comment as in outcome 4, analysis 11]; p < 0.001, cLDA model; GMT Ratio = 3.30, 95% CI 2-sided [2.91 to 3.74] — V116/PCV20
Statistical Analysis 13: Comparison: Cohort 1 V116 vs Cohort 1 PCV20; Serotype 15C: V116/PCV20 GMT Ratio; Test type: Superiority — [test comment as in outcome 4, analysis 11]; p < 0.001, cLDA model; GMT Ratio = 2.03, 95% CI 2-sided [1.77 to 2.34] — V116/PCV20
Statistical Analysis 14: Comparison: Cohort 1 V116 vs Cohort 1 PCV20; Serotype 16F: V116/PCV20 GMT Ratio; Test type: Superiority — [test comment as in outcome 4, analysis 11]; p < 0.001, cLDA model; GMT Ratio = 5.75, 95% CI 2-sided [5.16 to 6.41] — V116/PCV20
Statistical Analysis 15: Comparison: Cohort 1 V116 vs Cohort 1 PCV20; Serotype 17F: V116/PCV20 GMT Ratio; Test type: Superiority — [test comment as in outcome 4, analysis 11]; p < 0.001, cLDA model; GMT Ratio = 16.86, 95% CI 2-sided [14.90 to 19.09] — V116/PCV20
Statistical Analysis 16: Comparison: Cohort 1 V116 vs Cohort 1 PCV20; Serotype 20A: V116/PCV20 GMT Ratio; Test type: Superiority — [test comment as in outcome 4, analysis 11]; p < 0.001, cLDA model; GMT Ratio = 9.66, 95% CI 2-sided [8.66 to 10.79] — V116/PCV20
Statistical Analysis 17: Comparison: Cohort 1 V116 vs Cohort 1 PCV20; Serotype 23A: V116/PCV20 GMT Ratio; Test type: Superiority — [test comment as in outcome 4, analysis 11]; p < 0.001, cLDA model; GMT Ratio = 8.10, 95% CI 2-sided [6.86 to 9.55] — V116/PCV20
Statistical Analysis 18: Comparison: Cohort 1 V116 vs Cohort 1 PCV20; Serotype 23B: V116/PCV20 GMT Ratio; Test type: Superiority — [test comment as in outcome 4, analysis 11]; p < 0.001, cLDA model; GMT Ratio = 10.09, 95% CI 2-sided [8.48 to 12.00] — V116/PCV20
Statistical Analysis 19: Comparison: Cohort 1 V116 vs Cohort 1 PCV20; Serotype 24F: V116/PCV20 GMT Ratio; Test type: Superiority — [test comment as in outcome 4, analysis 11]; p < 0.001, cLDA model; GMT Ratio = 38.71, 95% CI 2-sided [33.87 to 44.25] — V116/PCV20
Statistical Analysis 20: Comparison: Cohort 1 V116 vs Cohort 1 PCV20; Serotype 31: V116/PCV20 GMT Ratio; Test type: Superiority — [test comment as in outcome 4, analysis 11]; p < 0.001, cLDA model; GMT Ratio = 21.69, 95% CI 2-sided [18.68 to 25.18] — V116/PCV20
Statistical Analysis 21: Comparison: Cohort 1 V116 vs Cohort 1 PCV20; Serotype 35B: V116/PCV20 GMT Ratio; Test type: Superiority — [test comment as in outcome 4, analysis 11]; p < 0.001, cLDA model; GMT Ratio = 6.17, 95% CI 2-sided [5.59 to 6.80] — V116/PCV20

5. Primary Outcome: Percentage of Participants With ≥4-fold Change From Baseline in Serotype Specific OPA Responses in Cohort 1 Only for the 11 Unique Pneumococcal Serotypes Contained in V116
Description: The percentage of participants with ≥4-fold rise from baseline in serotype specific OPAs for the 11 unique pneumococcal serotypes contained in V116. Per protocol, within group CIs or any other measures of dispersion were not planned or determined. The 11 unique pneumococcal serotypes in V116 were as follows: 9N, 15A, 15C, 16F, 17F, 20A, 23A, 23B, 24F, 31, and 35B. Per protocol, Cohort 2 were not analyzed in this outcome measure.
Time Frame: Baseline and Day 30 post-vaccination
Population: All randomized participants from cohort 1 only, without deviations from the protocol that may substantially affect immunogenicity. Deviations include, but are not limited to the following: missing serology results; and blood draw out of window. Cohort 2 were not analyzed in this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1 V116 | Cohort 1 PCV20 | Cohort 2 V116 | Cohort 2 PCV20
Number analyzed (Participants) | 1179 | 1177 | 0 | 0
Percentage of participants
  Serotype 9N: number analyzed (Participants) | 920 | 978 | 0 | 0
  Serotype 9N | 64.7 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 19.9 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 15A: number analyzed (Participants) | 693 | 706 | 0 | 0
  Serotype 15A | 66.7 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 35.8 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 15C: number analyzed (Participants) | 952 | 937 | 0 | 0
  Serotype 15C | 83.4 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 74.2 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 16F: number analyzed (Participants) | 910 | 961 | 0 | 0
  Serotype 16F | 71.9 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 20.8 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 17F: number analyzed (Participants) | 862 | 952 | 0 | 0
  Serotype 17F | 75.8 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 9.5 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 20A: number analyzed (Participants) | 1003 | 1011 | 0 | 0
  Serotype 20A | 67.3 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 9.6 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 23A: number analyzed (Participants) | 758 | 734 | 0 | 0
  Serotype 23A | 78.9 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 36.8 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 23B: number analyzed (Participants) | 1021 | 1021 | 0 | 0
  Serotype 23B | 85.5 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 49.6 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 24F: number analyzed (Participants) | 925 | 872 | 0 | 0
  Serotype 24F | 80.5 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 6.3 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 31: number analyzed (Participants) | 912 | 954 | 0 | 0
  Serotype 31 | 76.5 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 17.9 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 35B: number analyzed (Participants) | 917 | 988 | 0 | 0
  Serotype 35B | 60.0 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 6.8 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
Statistical Analysis 1: Comparison: Cohort 1 V116 vs Cohort 1 PCV20; Serotype 9N: V116-PCV20 Percentage Difference; Test type: Superiority — A conclusion of superiority is based on the lower bound of the 95% CI for the difference [V116 - PCV20] between the percentages of participants with a ≥4-fold rise from baseline being >10 percentage points (one-sided p-value < 0.025); p < 0.001, Stratified Miettinen & Nurminen — 1-sided; Percent Difference = 44.7, 95% CI 2-sided [40.7 to 48.6] — V116 minus PCV20
Statistical Analysis 2: Comparison: Cohort 1 V116 vs Cohort 1 PCV20; Serotype 15A: V116-PCV20 Percentage Difference; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p < 0.001, Stratified Miettinen & Nurminen — 1-sided; Percent Difference = 30.9, 95% CI 2-sided [25.8 to 35.8] — V116 minus PCV20
Statistical Analysis 3: Comparison: Cohort 1 V116 vs Cohort 1 PCV20; Serotype 15C: V116-PCV20 Percentage Difference; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p < 0.001, Stratified Miettinen & Nurminen — 1-sided; Percent Difference = 9.2, 95% CI 2-sided [5.6 to 12.9] — V116 minus PCV20
Statistical Analysis 4: Comparison: Cohort 1 V116 vs Cohort 1 PCV20; Serotype 16F: V116-PCV20 Percentage Difference; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p < 0.001, Stratified Miettinen & Nurminen — 1-sided; Percent Difference = 51.1, 95% CI 2-sided [47.1 to 54.9] — V116 minus PCV20
Statistical Analysis 5: Comparison: Cohort 1 V116 vs Cohort 1 PCV20; Serotype 17F: V116-PCV20 Percentage Difference; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p < 0.001, Stratified Miettinen & Nurminen — 1-sided; Percent Difference = 66.3, 95% CI 2-sided [62.8 to 69.6] — V116 minus PCV20
Statistical Analysis 6: Comparison: Cohort 1 V116 vs Cohort 1 PCV20; Serotype 20A: V116-PCV20 Percentage Difference; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p < 0.001, Stratified Miettinen & Nurminen — 1-sided; Percent Difference = 57.7, 95% CI 2-sided [54.2 to 61.1] — V116 minus PCV20
Statistical Analysis 7: Comparison: Cohort 1 V116 vs Cohort 1 PCV20; Serotype 23A: V116-PCV20 Percentage Difference; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p < 0.001, Stratified Miettinen & Nurminen — 1-sided; Percent Difference = 42.2, 95% CI 2-sided [37.6 to 46.6] — V116 minus PCV20
Statistical Analysis 8: Comparison: Cohort 1 V116 vs Cohort 1 PCV20; Serotype 23B: V116-PCV20 Percentage Difference; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p < 0.001, Stratified Miettinen & Nurminen — 1-sided; Percent Difference = 35.9, 95% CI 2-sided [32.1 to 39.6] — V116 minus PCV20
Statistical Analysis 9: Comparison: Cohort 1 V116 vs Cohort 1 PCV20; Serotype24F: V116-PCV20 Percentage Difference; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p < 0.001, Stratified Miettinen & Nurminen — 1-sided; Percent Difference = 74.2, 95% CI 2-sided [71.1 to 77.1] — V116 minus PCV20
Statistical Analysis 10: Comparison: Cohort 1 V116 vs Cohort 1 PCV20; Serotype 31: V116-PCV20 Percentage Difference; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p < 0.001, Stratified Miettinen & Nurminen — 1-sided; Percent Difference = 58.6, 95% CI 2-sided [54.8 to 62.1] — V116 minus PCV20
Statistical Analysis 11: Comparison: Cohort 1 V116 vs Cohort 1 PCV20; Serotype35B: V116-PCV20 Percentage Difference; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p < 0.001, Stratified Miettinen & Nurminen — 1-sided; Percent Difference = 53.2, 95% CI 2-sided [49.6 to 56.6] — V116 minus PCV20

6. Primary Outcome: Serotype Specific OPA GMTs in Participants 18-49 Years and Participants 50-64 Years for the Pneumococcal Serotypes Contained in V116
Description: The serotype specific OPA GMTs for the pneumococcal serotypes in participants 18-49 years and participants 50-64 years treated with V116 only were determined using the MOPA. GMT values were estimated from a cLDA model. Per protocol, within group CIs or any other measures of dispersion were not planned or determined. The 10 common pneumococcal serotypes in both V116 and PCV20 were as follows: 3, 6A, 7F, 8, 10A, 11A, 12F, 19A, 22F, and 33F. The 11 unique pneumococcal serotypes in V116 were as follows: 9N, 15A, 15C, 16F, 17F, 20A, 23A, 23B, 24F, 31, and 35B. Per protocol, participants treated with PCV20 were not analyzed in this outcome measure.
Time Frame: Day 30 post-vaccination
Population: All randomized participants treated with V116 only, without deviations from the protocol that may substantially affect immunogenicity. Deviations include, but are not limited to the following: missing serology results; and blood draw out of window. Per protocol, participants treated with PCV20 were not analyzed in this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Groups:
- V116 18 to 49 Years Old: Pneumococcal vaccine-naïve adult participants 18 to 49 years of age receive a single dose of V116 on Day 1.
- V116 50 to 64 Years Old: Pneumococcal vaccine-naïve adult participants 50 to 64 years of age receive a single dose of V116 on Day 1.
Arm/Group | V116 18 to 49 Years Old | V116 50 to 64 Years Old | Cohort 1 PCV20 | Cohort 2 PCV20
Number analyzed (Participants) | 200 | 589 | 0 | 0
Titer
  Serotype 3: number analyzed (Participants) | 194 | 572 | 0 | 0
  Serotype 3 | 308.6 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 282.7 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 6A: number analyzed (Participants) | 196 | 569 | 0 | 0
  Serotype 6A | 5289.6 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 2572.9 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 7F: number analyzed (Participants) | 198 | 571 | 0 | 0
  Serotype 7F | 6447.2 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 4278.8 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 8: number analyzed (Participants) | 197 | 571 | 0 | 0
  Serotype 8 | 4516.0 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 3004.7 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 9N: number analyzed (Participants) | 197 | 570 | 0 | 0
  Serotype 9N | 17283.2 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 8791.4 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 10A: number analyzed (Participants) | 197 | 575 | 0 | 0
  Serotype 10A | 6808.1 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 4382.6 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 11A: number analyzed (Participants) | 196 | 564 | 0 | 0
  Serotype 11A | 5871.6 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 3785.8 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 12F: number analyzed (Participants) | 196 | 574 | 0 | 0
  Serotype 12F | 6150.4 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 3561.2 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 15A: number analyzed (Participants) | 184 | 550 | 0 | 0
  Serotype 15A | 11319.2 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 5901.2 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 15C: number analyzed (Participants) | 195 | 570 | 0 | 0
  Serotype 15C | 10194.0 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 5708.0 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 16F: number analyzed (Participants) | 193 | 571 | 0 | 0
  Serotype 16F | 8877.0 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 5720.0 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype17F: number analyzed (Participants) | 194 | 568 | 0 | 0
  Serotype17F | 16070.6 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 10068.0 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 19A: number analyzed (Participants) | 198 | 574 | 0 | 0
  Serotype 19A | 2773.2 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 2374.6 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 20A: number analyzed (Participants) | 197 | 575 | 0 | 0
  Serotype 20A | 13150.0 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 7562.7 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 22F: number analyzed (Participants) | 198 | 568 | 0 | 0
  Serotype 22F | 9299.6 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 4683.6 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 23A: number analyzed (Participants) | 192 | 561 | 0 | 0
  Serotype 23A | 8848.7 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 4739.5 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 23B: number analyzed (Participants) | 198 | 575 | 0 | 0
  Serotype 23B | 2140.1 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 1420.9 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 24F: number analyzed (Participants) | 197 | 570 | 0 | 0
  Serotype 24F | 4137.6 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 3047.2 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 31: number analyzed (Participants) | 195 | 570 | 0 | 0
  Serotype 31 | 8005.6 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 3820.7 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 33F: number analyzed (Participants) | 197 | 570 | 0 | 0
  Serotype 33F | 34805.5 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 17607.4 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 35B: number analyzed (Participants) | 198 | 573 | 0 | 0
  Serotype 35B | 13933.4 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 9053.9 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
Statistical Analysis 1: Comparison: V116 18 to 49 Years Old vs V116 50 to 64 Years Old; Serotype 3: V116 18-49 years/V116 50-64 years GMT Ratio; Test type: Other — A conclusion of immunobridging is based on the lower bound of the 95% CI for the estimated GMT ratio (V116 18-49 Years/V116 50-64 Years) being > 0.5 (one-sided p-value < 0.025); p < 0.001, LDA model — 1-sided; GMT Ratio = 1.09, 95% CI 2-sided [0.90 to 1.33] — V116 18-49 years/V116 50-64 years
Statistical Analysis 2: Comparison: V116 18 to 49 Years Old vs V116 50 to 64 Years Old; Serotype 6A: V116 18-49 years/V116 50-64 years GMT Ratio; Test type: Other — [test comment as in outcome 6, analysis 1]; p < 0.001, LDA model — 1-sided; GMT Ratio = 2.06, 95% CI 2-sided [1.61 to 2.62] — V116 18-49 years/V116 50-64 years
Statistical Analysis 3: Comparison: V116 18 to 49 Years Old vs V116 50 to 64 Years Old; Serotype 7F: V116 18-49 years/V116 50-64 years GMT Ratio; Test type: Other — [test comment as in outcome 6, analysis 1]; p < 0.001, LDA model — 1-sided; GMT Ratio = 1.51, 05% CI 2-sided [1.23 to 1.84] — V116 18-49 years/V116 50-64 years
Statistical Analysis 4: Comparison: V116 18 to 49 Years Old vs V116 50 to 64 Years Old; Serotype 8: V116 18-49 years/V116 50-64 years GMT Ratio; Test type: Other — [test comment as in outcome 6, analysis 1]; p < 0.001, LDA model — 1-sided; GMT Ratio = 1.50, 95% CI 2-sided [1.26 to 1.79] — V116 18-49 years/V116 50-64 years
Statistical Analysis 5: Comparison: V116 18 to 49 Years Old vs V116 50 to 64 Years Old; Serotype 9N: V116 18-49 years/V116 50-64 years GMT Ratio; Test type: Other — [test comment as in outcome 6, analysis 1]; p < 0.001, LDA model — 1-sided; GMT Ratio = 1.97, 95% CI 2-sided [1.59 to 2.43] — V116 18-49 years/V116 50-64 years
Statistical Analysis 6: Comparison: V116 18 to 49 Years Old vs V116 50 to 64 Years Old; Serotype 10A: V116 18-49 years/V116 50-64 years GMT Ratio; Test type: Other — [test comment as in outcome 6, analysis 1]; p < 0.001, LDA model — 1-sided; GMT Ratio = 1.55, 95% CI 2-sided [1.26 to 1.92] — V116 18-49 years/V116 50-64 years
Statistical Analysis 7: Comparison: V116 18 to 49 Years Old vs V116 50 to 64 Years Old; Serotype 11A: V116 18-49 years/V116 50-64 years GMT Ratio; Test type: Other — [test comment as in outcome 6, analysis 1]; p < 0.001, LDA model — 1-sided; GMT Ratio = 1.55, 95% CI 2-sided [1.26 to 1.91] — V116 18-49 years/V116 50-64 years
Statistical Analysis 8: Comparison: V116 18 to 49 Years Old vs V116 50 to 64 Years Old; Serotype 12F: V116 18-49 years/V116 50-64 years GMT Ratio; Test type: Other — [test comment as in outcome 6, analysis 1]; p < 0.001, LDA model — 1-sided; GMT Ratio = 1.73, 95% CI 2-sided [1.37 to 2.17] — V116 18-49 years/V116 50-64 years
Statistical Analysis 9: Comparison: V116 18 to 49 Years Old vs V116 50 to 64 Years Old; Serotype 15A: V116 18-49 years/V116 50-64 years GMT Ratio; Test type: Other — [test comment as in outcome 6, analysis 1]; p < 0.001, LDA model — 1-sided; GMT Ratio = 1.92, 95% CI 2-sided [1.55 to 2.37] — V116 18-49 years/V116 50-64 years
Statistical Analysis 10: Comparison: V116 18 to 49 Years Old vs V116 50 to 64 Years Old; Serotype 15C: V116 18-49 years/V116 50-64 years GMT Ratio; Test type: Other — [test comment as in outcome 6, analysis 1]; p < 0.001, LDA model — 1-sided; GMT Ratio = 1.79, 95% CI 2-sided [1.36 to 2.35] — V116 18-49 years/V116 50-64 years
Statistical Analysis 11: Comparison: V116 18 to 49 Years Old vs V116 50 to 64 Years Old; Serotype 16F: V116 18-49 years/V116 50-64 years GMT Ratio; Test type: Other — [test comment as in outcome 6, analysis 1]; p < 0.001, LDA model — 1-sided; GMT Ratio = 1.55, 95% CI 2-sided [1.26 to 1.91] — V116 18-49 years/V116 50-64 years
Statistical Analysis 12: Comparison: V116 18 to 49 Years Old vs V116 50 to 64 Years Old; Serotype 17F: V116 18-49 years/V116 50-64 years GMT Ratio; Test type: Other — [test comment as in outcome 6, analysis 1]; p < 0.001, LDA model — 1-sided; GMT Ratio = 1.60, 95% CI 2-sided [1.26 to 2.02] — V116 18-49 years/V116 50-64 years
Statistical Analysis 13: Comparison: V116 18 to 49 Years Old vs V116 50 to 64 Years Old; Serotype 19A: V116 18-49 years/V116 50-64 years GMT Ratio; Test type: Other — [test comment as in outcome 6, analysis 1]; p < 0.001, LDA model — 1-sided; GMT Ratio = 1.17, 95% CI 2-sided [0.97 to 1.40] — V116 18-49 years/V116 50-64 years
Statistical Analysis 14: Comparison: V116 18 to 49 Years Old vs V116 50 to 64 Years Old; Serotype 20A: V116 18-49 years/V116 50-64 years GMT Ratio; Test type: Other — [test comment as in outcome 6, analysis 1]; p < 0.001, LDA model — 1-sided; GMT Ratio = 1.74, 95% CI 2-sided [1.39 to 2.18] — V116 18-49 years/V116 50-64 years
Statistical Analysis 15: Comparison: V116 18 to 49 Years Old vs V116 50 to 64 Years Old; Serotype 22F: V116 18-49 years/V116 50-64 years GMT Ratio; Test type: Other — [test comment as in outcome 6, analysis 1]; p < 0.001, LDA model — 1-sided; GMT Ratio = 1.99, 95% CI 2-sided [1.58 to 2.49] — V116 18-49 years/V116 50-64 years
Statistical Analysis 16: Comparison: V116 18 to 49 Years Old vs V116 50 to 64 Years Old; Serotype 23A: V116 18-49 years/V116 50-64 years GMT Ratio; Test type: Other — [test comment as in outcome 6, analysis 1]; p < 0.001, LDA model — 1-sided; GMT Ratio = 1.87, 95% CI 2-sided [1.43 to 2.44] — V116 18-49 years/V116 50-64 years
Statistical Analysis 17: Comparison: V116 18 to 49 Years Old vs V116 50 to 64 Years Old; Serotype 23B: V116 18-49 years/V116 50-64 years GMT Ratio; Test type: Other — [test comment as in outcome 6, analysis 1]; p < 0.001, LDA model — 1-sided; GMT Ratio = 1.51, 95% CI 2-sided [1.11 to 2.04] — V116 18-49 years/V116 50-64 years
Statistical Analysis 18: Comparison: V116 18 to 49 Years Old vs V116 50 to 64 Years Old; Serotype 24F: V116 18-49 years/V116 50-64 years GMT Ratio; Test type: Other — [test comment as in outcome 6, analysis 1]; p < 0.001, LDA model — 1-sided; GMT Ratio = 1.36, 95% CI 2-sided [1.10 to 1.67] — V116 18-49 years/V116 50-64 years
Statistical Analysis 19: Comparison: V116 18 to 49 Years Old vs V116 50 to 64 Years Old; Serotype 31: V116 18-49 years/V116 50-64 years GMT Ratio; Test type: Other — [test comment as in outcome 6, analysis 1]; p < 0.001, LDA model — 1-sided; GMT Ratio = 2.10, 95% CI 2-sided [1.63 to 2.69] — V116 18-49 years/V116 50-64 years
Statistical Analysis 20: Comparison: V116 18 to 49 Years Old vs V116 50 to 64 Years Old; Serotype 33F: V116 18-49 years/V116 50-64 years GMT Ratio; Test type: Other — [test comment as in outcome 6, analysis 1]; p < 0.001, LDA model — 1-sided; GMT Ratio = 1.98, 95% CI 2-sided [1.52 to 2.57] — V116 18-49 years/V116 50-64 years
Statistical Analysis 21: Comparison: V116 18 to 49 Years Old vs V116 50 to 64 Years Old; Serotype 35B: V116 18-49 years/V116 50-64 years GMT Ratio; Test type: Other — [test comment as in outcome 6, analysis 1]; p < 0.001, LDA model — 1-sided; GMT Ratio = 1.54, 95% CI 2-sided [1.26 to 1.87] — V116 18-49 years/V116 50-64 years

7. Secondary Outcome: Percentage of Participants From Cohort 1 V116 With ≥4-fold Change in OPA Responses for Cross Reactive Pneumococcal Serotypes
Description: The percentage of participants with ≥4-fold rise from baseline was determined for Cohort 1 V116 serotypes 6C and 15B, two serotypes which cross react with PCV20. Point estimate and 95% CI are based on the Clopper-Pearson method. A conclusion of acceptability is based on the lower bound of the 95% CI of the percentages of participants with a ≥4-fold rise from baseline being > 50 percentage points (one-sided p-value < 0.025). Per protocol, participants treated with PCV20, and V116 Cohort 2 were not analyzed in this outcome measure.
Time Frame: Baseline and Day 30 post-vaccination
Population: All randomized participants treated with V116 only, without deviations from the protocol that may substantially affect immunogenicity. Deviations include, but are not limited to the following: missing serology results; and blood draw out of window. Per protocol, participants treated with PCV20 and V116 Cohort 2 were not analyzed in this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1 V116 | Cohort 1 PCV20 | Cohort 2 V116 | Cohort 2 PCV20
Number analyzed (Participants) | 1179 | 0 | 0 | 0
Percentage of participants
  Serotype 6C: number analyzed (Participants) | 912 | 0 | 0 | 0
  Serotype 6C | 49.3 [46.0 to 52.6] |  |  |
  Serotype 15B: number analyzed (Participants) | 883 | 0 | 0 | 0
  Serotype 15B | 64.7 [61.4 to 67.8] |  |  |
Statistical Analysis 1: Comparison: Cohort 1 V116; Serotype 6C; Test type: Other — A conclusion of acceptability is based on the lower bound of the 95% CI of the percentages of participants with a ≥4-fold rise from baseline to 30 days postvaccination being > 50 percentage points (one-sided p-value < 0.025); p = 0.667, Clopper-Pearson method. — 1-sided
Statistical Analysis 2: Comparison: Cohort 1 V116; Serotype 15B; Test type: Other — [test comment as in outcome 7, analysis 1]; p < 0.001, Clopper-Pearson method. — 1-sided

8. Secondary Outcome: Serotype Specific OPA GMTs for Cross Reactive Pneumococcal Serotypes in Adults 50 to 64 Years of Age From Cohort 1 and Adults 18 to 49 Years of Age From Cohort 2
Description: The serotype specific OPA GMTs for the pneumococcal serotypes in participants 18-49 years and participants 50-64 years treated with V116 only were determined using the MOPA for serotypes 6C and 15B which cross react with PCV20. GMT values were estimated from a LDA model. Per protocol, within group CIs or any other measures of dispersion were not planned or determined. Per protocol, participants treated with PCV20 were not analyzed in this outcome measure.
Time Frame: Day 30 post-vaccination
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Groups:
- V116 18 to 49 Years Old: Pneumococcal vaccine-naïve adult participants in Cohort 2 (18 to 49 years of age) receive a single dose of V116 on Day 1.
- V116 50 to 64 Years Old: Pneumococcal vaccine-naïve adult participants n Cohort 1 50 to 64 years of age receive a single dose of V116 on Day 1.
Arm/Group | V116 18 to 49 Years Old | V116 50 to 64 Years Old | Cohort 1 PCV20 | Cohort 2 PCV20
Number analyzed (Participants) | 200 | 589 | 0 | 0
Titer
  6C: number analyzed (Participants) | 194 | 570 | 0 | 0
  6C | 2577.2 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 1254.7 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  15B: number analyzed (Participants) | 192 | 566 | 0 | 0
  15B | 10976.7 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 5438.9 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
Statistical Analysis 1: Comparison: V116 18 to 49 Years Old vs V116 50 to 64 Years Old; Serotype 6C: V116 18-49 years/V116 50-64 years GMT Ratio; Test type: Other — [test comment as in outcome 6, analysis 1]; GMT Ratio = 2.05, 95% CI 2-sided [1.52 to 2.77] — V116 18-49 years/V116 50-64 years
Statistical Analysis 2: Comparison: V116 18 to 49 Years Old vs V116 50 to 64 Years Old; Serotype 15B: V116 18-49 years/V116 50-64 years GMT ratio; Test type: Other — [test comment as in outcome 6, analysis 1]; p < 0.001, LDA model — 1-sided; GMT = 2.02, 95% CI 2-sided [1.57 to 2.60] — V116 18-49 years/V116 50-64 years

9. Secondary Outcome: Serotype Specific Immunoglobulin (IgG) Geometric Mean Concentrations (GMCs) in Cohort 1 Only, for the Pneumococcal Serotypes Contained in V116 and PCV20
Description: The serotype specific IgG GMCs for the pneumococcal serotypes in cohort 1 of V116 and PCV20 only were determined using pneumococcal electrochemiluminescence (PnECL). GMC values were estimated from a cLDA model. Per protocol, within group CIs or any other measures of dispersion were not planned or determined. The 10 common pneumococcal serotypes in both V116 and PCV20 were as follows: 3, 6A, 7F, 8, 10A, 11A, 12F, 19A, 22F, and 33F. The 11 unique pneumococcal serotypes in V116 were as follows: 9N, 15A, 15C, 16F, 17F, 20A, 23A, 23B, 24F, 31, and 35B. Per protocol, Cohort 2 were not analyzed in this outcome measure.
Time Frame: Day 30 post-vaccination
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Cohort 1 V116 | Cohort 1 PCV20 | Cohort 2 V116 | Cohort 2 PCV20
Number analyzed (Participants) | 1179 | 1177 | 0 | 0
μg/mL
  Serotype 3: number analyzed (Participants) | 1166 | 1167 | 0 | 0
  Serotype 3 | 0.78 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 0.53 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 6A: number analyzed (Participants) | 1166 | 1167 | 0 | 0
  Serotype 6A | 4.30 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 5.45 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 7F: number analyzed (Participants) | 1166 | 1167 | 0 | 0
  Serotype 7F | 6.97 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 6.57 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 8: number analyzed (Participants) | 1166 | 1167 | 0 | 0
  Serotype 8 | 10.02 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 7.00 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 10A: number analyzed (Participants) | 1166 | 1167 | 0 | 0
  Serotype 10A | 11.98 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 14.66 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 11A: number analyzed (Participants) | 1166 | 1167 | 0 | 0
  Serotype 11A | 7.20 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 5.87 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 12F: number analyzed (Participants) | 1166 | 1167 | 0 | 0
  Serotype 12F | 1.73 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 1.57 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 19A: number analyzed (Participants) | 1166 | 1167 | 0 | 0
  Serotype 19A | 8.39 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 12.02 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 22F: number analyzed (Participants) | 1166 | 1167 | 0 | 0
  Serotype 22F | 4.39 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 5.48 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 33F: number analyzed (Participants) | 1166 | 1167 | 0 | 0
  Serotype 33F | 13.81 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 13.02 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined.. |  |
  Serotype 9N: number analyzed (Participants) | 1166 | 1167 | 0 | 0
  Serotype 9N | 7.72 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 1.43 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype15A: number analyzed (Participants) | 1166 | 1167 | 0 | 0
  Serotype15A | 13.88 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 2.04 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 15C: number analyzed (Participants) | 1166 | 1167 | 0 | 0
  Serotype 15C | 12.39 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 5.04 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 16F: number analyzed (Participants) | 1166 | 1167 | 0 | 0
  Serotype 16F | 2.86 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 0.33 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 17F: number analyzed (Participants) | 1166 | 1167 | 0 | 0
  Serotype 17F | 14.16 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 0.84 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 20A: number analyzed (Participants) | 1166 | 1167 | 0 | 0
  Serotype 20A | 19.03 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 1.47 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 23A: number analyzed (Participants) | 1166 | 1167 | 0 | 0
  Serotype 23A | 3.78 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 0.59 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 23B: number analyzed (Participants) | 1166 | 1167 | 0 | 0
  Serotype 23B | 5.13 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 1.58 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 24F: number analyzed (Participants) | 1166 | 1167 | 0 | 0
  Serotype 24F | 6.87 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 0.33 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 31: number analyzed (Participants) | 1166 | 1167 | 0 | 0
  Serotype 31 | 3.07 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 0.27 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
  Serotype 35B: number analyzed (Participants) | 1166 | 1167 | 0 | 0
  Serotype 35B | 19.98 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. | 1.41 [NA to NA] — NA: per protocol, within group CIs, or any other measures of dispersion, were not determined. |  |
Statistical Analysis 1: Comparison: Cohort 1 V116 vs Cohort 1 PCV20; Serotype 3: V116/PCV20 GMC Ratio; Test type: Other — cLDA model; GMC Ratio = 1.47, 95% CI 2-sided [1.35 to 1.60] — V116/PCV20
Statistical Analysis 2: Comparison: Cohort 1 V116 vs Cohort 1 PCV20; Serotype 6A: V116/PCV20 GMC Ratio; Test type: Other — cLDA model; GMC Ratio = 0.79, 95% CI 2-sided [0.70 to 0.89] — V116/PCV20
Statistical Analysis 3: Comparison: Cohort 1 V116 vs Cohort 1 PCV20; Serotype 7F: V116/PCV20 GMC Ratio; Test type: Other — cLDA model; GMC Ratio = 1.06, 95% CI 2-sided [0.95 to 1.18] — V116/PCV20
Statistical Analysis 4: Comparison: Cohort 1 V116 vs Cohort 1 PCV20; Serotype 8: V116/PCV20 GMC Ratio; Test type: Other — cLDA model; GMC Ratio = 1.43, 95% CI 2-sided [1.29 to 1.59] — V116/PCV20
Statistical Analysis 5: Comparison: Cohort 1 V116 vs Cohort 1 PCV20; Serotype 10A: V116/PCV20 GMC Ratio; Test type: Other — cLDA model; GMC Ratio = 0.82, 95% CI 2-sided [0.72 to 0.92] — V116/PCV20
Statistical Analysis 6: Comparison: Cohort 1 V116 vs Cohort 1 PCV20; Serotype 11A: V116/PCV20 GMC Ratio; Test type: Other — cLDA model; GMC Ratio = 1.23, 95% CI 2-sided [1.11 to 1.36] — V116/PCV20
Statistical Analysis 7: Comparison: Cohort 1 V116 vs Cohort 1 PCV20; Serotype 12F: V116/PCV20 GMC Ratio; Test type: Other — cLDA model; GMC Ratio = 1.10, 95% CI 2-sided [0.96 to 1.26] — V116/PCV20
Statistical Analysis 8: Comparison: Cohort 1 V116 vs Cohort 1 PCV20; Serotype 19A: V116/PCV20 GMC Ratio; Test type: Other — cLDA model; GMC Ratio = 0.70, 95% CI 2-sided [0.63 to 0.77] — V116/PCV20
Statistical Analysis 9: Comparison: Cohort 1 V116 vs Cohort 1 PCV20; Serotype 22F: V116/PCV20 GMC Ratio; Test type: Other — cLDA model; GMC Ratio = 0.80, 95% CI 2-sided [0.72 to 0.90] — V116/PCV20
Statistical Analysis 10: Comparison: Cohort 1 V116 vs Cohort 1 PCV20; Serotype 33F: V116/PCV20 GMC Ratio; Test type: Other — cLDA model; GMC Ratio = 1.06, 95% CI 2-sided [0.95 to 1.18] — V116/PCV20
Statistical Analysis 11: Comparison: Cohort 1 V116 vs Cohort 1 PCV20; Serotype 9N: V116/PCV20 GMC Ratio; Test type: Other — cLDA model; GMC Ratio = 5.41, 95% CI 2-sided [4.82 to 6.06] — V116/PCV20
Statistical Analysis 12: Comparison: Cohort 1 V116 vs Cohort 1 PCV20; Serotype 15A: V116/PCV20 GMC Ratio; Test type: Other — cLDA model; GMC Ratio = 6.79, 95% CI 2-sided [6.03 to 7.64] — V116/PCV20
Statistical Analysis 13: Comparison: Cohort 1 V116 vs Cohort 1 PCV20; Serotype 15C: V116/PCV20 GMC Ratio; Test type: Other — cLDA model; GMC Ratio = 2.46, 95% CI 2-sided [2.17 to 2.79] — V116/PCV20
Statistical Analysis 14: Comparison: Cohort 1 V116 vs Cohort 1 PCV20; Serotype 16F: V116/PCV20 GMC Ratio; Test type: Other — cLDA model; GMC Ratio = 8.75, 95% CI 2-sided [7.95 to 9.64] — V116/PCV20
Statistical Analysis 15: Comparison: Cohort 1 V116 vs Cohort 1 PCV20; Serotype 17F: V116/PCV20 GMC Ratio; Test type: Other — cLDA model; GMC Ratio = 16.75, 95% CI 2-sided [15.25 to 18.41] — V116/PCV20
Statistical Analysis 16: Comparison: Cohort 1 V116 vs Cohort 1 PCV20; Serotype 20A: V116/PCV20 GMC Ratio; Test type: Other — cLDA model; GMC Ratio = 12.92, 05% CI 2-sided [11.81 to 14.13] — V116/PCV20
Statistical Analysis 17: Comparison: Cohort 1 V116 vs Cohort 1 PCV20; Serotype 23A: V116/PCV20 GMC Ratio; Test type: Other — cLDA model; GMC Ratio = 6.42, 95% CI 2-sided [5.69 to 7.24] — V116/PCV20
Statistical Analysis 18: Comparison: Cohort 1 V116 vs Cohort 1 PCV20; Serotype 23B: V116/PCV20 GMC Ratio; Test type: Other — cLDA model; GMC Ratio = 3.25, 95% CI 2-sided [2.91 to 3.64] — V116/PCV20
Statistical Analysis 19: Comparison: Cohort 1 V116 vs Cohort 1 PCV20; Serotype 24F: V116/PCV20 GMC Ratio; Test type: Other — cLDA model; GMC Ratio = 21.08, 85% CI 2-sided [18.97 to 23.43] — V116/PCV20
Statistical Analysis 20: Comparison: Cohort 1 V116 vs Cohort 1 PCV20; Serotype 31: V116/PCV20 GMC Ratio; Test type: Other — cLDA model; GMC Ratio = 11.31, 95% CI 2-sided [10.36 to 12.34] — V116/PCV20
Statistical Analysis 21: Comparison: Cohort 1 V116 vs Cohort 1 PCV20; Serotype 35B: V116/PCV20 GMC Ratio; Test type: Other — cLDA model; GMC Ratio = 14.13, 95% CI 2-sided [12.97 to 15.40] — V116/PCV20

10. Secondary Outcome: Geometric Mean Fold Change From Baseline in OPA GMTs in Cohort 1 for the Pneumococcal Serotypes Contained in V116 and PCV20
Description: The geometric mean fold rise (GMFR) from baseline in serotype specific OPA GMTs for cohort 1 was determined using MOPA. The within-group 95% CIs were obtained by exponentiating the CIs of the mean of the natural log values based on the t-distribution. The 10 common pneumococcal serotypes in both V116 and PCV20 were as follows: 3, 6A, 7F, 8, 10A, 11A, 12F, 19A, 22F, and 33F. The 11 unique pneumococcal serotypes in V116 were as follows: 9N, 15A, 15C, 16F, 17F, 20A, 23A, 23B, 24F, 31, and 35B. Per protocol, Cohort 2 were not analyzed in this outcome measure.
Time Frame: Baseline and Day 30 post-vaccination
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: GMFR
Arm/Group | Cohort 1 V116 | Cohort 1 PCV20 | Cohort 2 V116 | Cohort 2 PCV20
Number analyzed (Participants) | 1179 | 1177 | 0 | 0
GMFR
  Serotype 3: number analyzed (Participants) | 966 | 937 | 0 | 0
  Serotype 3 | 8.4 [7.7 to 9.1] | 5.4 [5.0 to 5.8] |  |
  Serotype 6A: number analyzed (Participants) | 954 | 931 | 0 | 0
  Serotype 6A | 18.1 [16.2 to 20.2] | 22.6 [20.1 to 25.5] |  |
  Serotype 7F: number analyzed (Participants) | 967 | 961 | 0 | 0
  Serotype 7F | 16.5 [14.4 to 18.8] | 14.7 [12.9 to 16.8] |  |
  Serotype 8: number analyzed (Participants) | 999 | 971 | 0 | 0
  Serotype 8 | 22.0 [19.3 to 25.0] | 14.2 [12.5 to 16.2] |  |
  Serotype 10A: number analyzed (Participants) | 1021 | 978 | 0 | 0
  Serotype 10A | 16.7 [14.8 to 18.9] | 20.8 [18.3 to 23.8] |  |
  Serotype11A: number analyzed (Participants) | 890 | 889 | 0 | 0
  Serotype11A | 17.4 [15.1 to 20.0] | 11.6 [10.1 to 13.3] |  |
  Serotype 12F: number analyzed (Participants) | 1031 | 1022 | 0 | 0
  Serotype 12F | 77.4 [68.5 to 87.4] | 73.5 [64.8 to 83.4] |  |
  Serotype 19A: number analyzed (Participants) | 1024 | 990 | 0 | 0
  Serotype 19A | 8.6 [7.7 to 9.5] | 11.0 [9.9 to 12.2] |  |
  Serotype 22F: number analyzed (Participants) | 936 | 935 | 0 | 0
  Serotype 22F | 19.1 [16.6 to 22.1] | 25.5 [21.9 to 29.8] |  |
  Serotype 33F: number analyzed (Participants) | 937 | 938 | 0 | 0
  Serotype 33F | 9.9 [8.9 to 11.1] | 8.5 [7.6 to 9.5] |  |
  Serotype 9N: number analyzed (Participants) | 920 | 978 | 0 | 0
  Serotype 9N | 8.9 [8.0 to 9.9] | 2.0 [1.9 to 2.2] |  |
  Serotype 15A: number analyzed (Participants) | 693 | 706 | 0 | 0
  Serotype 15A | 9.4 [8.2 to 10.8] | 3.1 [2.7 to 3.5] |  |
  Serotype 15C: number analyzed (Participants) | 952 | 937 | 0 | 0
  Serotype 15C | 38.0 [33.3 to 43.3] | 20.3 [17.8 to 23.1] |  |
  Serotype 16F: number analyzed (Participants) | 910 | 961 | 0 | 0
  Serotype 16F | 9.5 [8.7 to 10.4] | 1.9 [1.7 to 2.0] |  |
  Serotype 17F: number analyzed (Participants) | 862 | 952 | 0 | 0
  Serotype 17F | 17.3 [15.3 to 19.7] | 1.2 [1.1 to 1.3] |  |
  Serotype 20A: number analyzed (Participants) | 1003 | 1011 | 0 | 0
  Serotype 20A | 10.3 [9.2 to 11.4] | 1.2 [1.1 to 1.2] |  |
  Serotype 23A: number analyzed (Participants) | 758 | 734 | 0 | 0
  Serotype 23A | 21.8 [19.0 to 25.0] | 3.1 [2.7 to 3.6] |  |
  Serotype 23B: number analyzed (Participants) | 1021 | 1021 | 0 | 0
  Serotype 23B | 51.4 [45.3 to 58.2] | 6.1 [5.4 to 6.9] |  |
  Serotype 24F: number analyzed (Participants) | 925 | 872 | 0 | 0
  Serotype 24F | 29.0 [25.6 to 32.8] | 1.1 [1.0 to 1.1] |  |
  Serotype 31: number analyzed (Participants) | 912 | 954 | 0 | 0
  Serotype 31 | 28.7 [24.9 to 33.1] | 1.5 [1.4 to 1.7] |  |
  Serotype 35B: number analyzed (Participants) | 917 | 988 | 0 | 0
  Serotype 35B | 7.2 [6.5 to 7.9] | 1.2 [1.1 to 1.2] |  |

11. Secondary Outcome: Geometric Mean Fold Change From Baseline in IgG Antibody GMCs in Cohort 1 for the Pneumococcal Serotypes Contained in V116 and PCV20
Description: The GMFR from baseline in serotype specific IgG antibody GMCs for cohort 1 was determined using PnECL. The within-group 95% CIs were obtained by exponentiating the CIs of the mean of the natural log values based on the t-distribution. The 10 common pneumococcal serotypes in both V116 and PCV20 were as follows: 3, 6A, 7F, 8, 10A, 11A, 12F, 19A, 22F, and 33F. The 11 unique pneumococcal serotypes in V116 were as follows: 9N, 15A, 15C, 16F, 17F, 20A, 23A, 23B, 24F, 31, and 35B. Per protocol, Cohort 2 were not analyzed in this outcome measure.
Time Frame: Baseline and Day 30 post-vaccination
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: GMFR
Arm/Group | Cohort 1 V116 | Cohort 1 PCV20 | Cohort 2 V116 | Cohort 2 PCV20
Number analyzed (Participants) | 1179 | 1177 | 0 | 0
GMFR
  Serotype 3: number analyzed (Participants) | 1101 | 1076 | 0 | 0
  Serotype 3 | 5.1 [4.8 to 5.4] | 3.5 [3.3 to 3.7] |  |
  Serotype 6A: number analyzed (Participants) | 1097 | 1069 | 0 | 0
  Serotype 6A | 12.2 [11.1 to 13.5] | 15.1 [13.8 to 16.6] |  |
  Serotype 7F: number analyzed (Participants) | 1097 | 1076 | 0 | 0
  Serotype 7F | 12.5 [11.5 to 13.7] | 12.2 [11.2 to 13.4] |  |
  Serotype 8: number analyzed (Participants) | 1102 | 1074 | 0 | 0
  Serotype 8 | 12.6 [11.5 to 13.8] | 8.8 [8.0 to 9.6] |  |
  Serotype 10A: number analyzed (Participants) | 1099 | 1070 | 0 | 0
  Serotype 10A | 15.4 [14.1 to 16.9] | 19.2 [17.4 to 21.1] |  |
  Serotype11A: number analyzed (Participants) | 1095 | 1071 | 0 | 0
  Serotype11A | 8.7 [8.1 to 9.5] | 7.1 [6.5 to 7.7] |  |
  Serotype 12F: number analyzed (Participants) | 1100 | 1073 | 0 | 0
  Serotype 12F | 13.1 [11.8 to 14.4] | 12.1 [11.0 to 13.5] |  |
  Serotype 19A: number analyzed (Participants) | 1098 | 1070 | 0 | 0
  Serotype 19A | 5.4 [5.0 to 5.8] | 7.7 [7.1 to 8.4] |  |
  Serotype 22F: number analyzed (Participants) | 1099 | 1076 | 0 | 0
  Serotype 22F | 12.7 [11.6 to 13.9] | 16.3 [14.8 to 17.9] |  |
  Serotype 33F: number analyzed (Participants) | 1097 | 1067 | 0 | 0
  Serotype 33F | 9.6 [8.8 to 10.5] | 9.1 [8.3 to 9.9] |  |
  Serotype 9N: number analyzed (Participants) | 1098 | 1074 | 0 | 0
  Serotype 9N | 15.0 [13.6 to 16.5] | 2.7 [2.5 to 2.9] |  |
  Serotype 15A: number analyzed (Participants) | 1087 | 1061 | 0 | 0
  Serotype 15A | 22.3 [20.3 to 24.4] | 3.4 [3.1 to 3.7] |  |
  Serotype 15C: number analyzed (Participants) | 1095 | 1071 | 0 | 0
  Serotype 15C | 19.8 [17.9 to 21.8] | 8.2 [7.4 to 9.0] |  |
  Serotype 16F: number analyzed (Participants) | 1090 | 1074 | 0 | 0
  Serotype 16F | 13.3 [12.3 to 14.4] | 1.6 [1.5 to 1.7] |  |
  Serotype 17F: number analyzed (Participants) | 1098 | 1076 | 0 | 0
  Serotype 17F | 19.8 [18.0 to 21.7] | 1.2 [1.1 to 1.3] |  |
  Serotype 20A: number analyzed (Participants) | 1097 | 1077 | 0 | 0
  Serotype 20A | 11.7 [10.8 to 12.8] | 0.9 [0.9 to 1.0] |  |
  Serotype 23A: number analyzed (Participants) | 1091 | 1074 | 0 | 0
  Serotype 23A | 17.8 [16.3 to 19.5] | 2.9 [2.6 to 3.1] |  |
  Serotype 23B: number analyzed (Participants) | 1094 | 1075 | 0 | 0
  Serotype 23B | 12.1 [11.1 to 13.3] | 3.8 [3.5 to 4.1] |  |
  Serotype 24F: number analyzed (Participants) | 1093 | 1077 | 0 | 0
  Serotype 24F | 21.2 [19.3 to 23.4] | 1.1 [1.0 to 1.1] |  |
  Serotype 31: number analyzed (Participants) | 1094 | 1075 | 0 | 0
  Serotype 31 | 13.0 [12.0 to 14.0] | 1.2 [1.2 to 1.3] |  |
  Serotype 35B: number analyzed (Participants) | 1090 | 1075 | 0 | 0
  Serotype 35B | 14.7 [13.6 to 16.0] | 1.0 [1.0 to 1.1] |  |

12. Secondary Outcome: Percentage of Participants With ≥4-fold Change From Baseline in IgG Antibody GMCs in Cohort 1 for the Pneumococcal Serotypes Contained in V116 and PCV20
Description: Percentage of participants with ≥4-fold rise from baseline in serotype specific IgG antibody GMCs for cohort 1 was determined using PnECL. The within-group 95% CIs were based on the exact binomial method proposed by Clopper and Pearson. The 10 common pneumococcal serotypes in both V116 and PCV20 were as follows: 3, 6A, 7F, 8, 10A, 11A, 12F, 19A, 22F, and 33F. The 11 unique pneumococcal serotypes in V116 were as follows: 9N, 15A, 15C, 16F, 17F, 20A, 23A, 23B, 24F, 31, and 35B. Per protocol, Cohort 2 were not analyzed in this outcome measure.
Time Frame: Baseline and Day 30 post-vaccination
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1 V116 | Cohort 1 PCV20 | Cohort 2 V116 | Cohort 2 PCV20
Number analyzed (Participants) | 1179 | 1177 | 0 | 0
Percentage of participants
  Serotype 3: number analyzed (Participants) | 1101 | 1076 | 0 | 0
  Serotype 3 | 56.5 [53.5 to 59.4] | 41.0 [38.0 to 44.0] |  |
  Serotype 6A: number analyzed (Participants) | 1097 | 1069 | 0 | 0
  Serotype 6A | 73.1 [70.4 to 75.7] | 79.7 [77.2 to 82.1] |  |
  Serotype 7F: number analyzed (Participants) | 1097 | 1076 | 0 | 0
  Serotype 7F | 76.4 [73.8 to 78.9] | 75.8 [73.2 to 78.4] |  |
  Serotype 8: number analyzed (Participants) | 1102 | 1074 | 0 | 0
  Serotype 8 | 75.8 [73.1 to 78.3] | 67.8 [64.9 to 70.6] |  |
  Serotype 10A: number analyzed (Participants) | 1099 | 1070 | 0 | 0
  Serotype 10A | 80.3 [77.8 to 82.6] | 82.0 [79.5 to 84.2] |  |
  Serotype11A: number analyzed (Participants) | 1095 | 1071 | 0 | 0
  Serotype11A | 71.1 [68.4 to 73.8] | 62.7 [59.8 to 65.6] |  |
  Serotype 12F: number analyzed (Participants) | 1100 | 1073 | 0 | 0
  Serotype 12F | 74.2 [71.5 to 76.7] | 71.4 [68.6 to 74.1] |  |
  Serotype 19A: number analyzed (Participants) | 1098 | 1070 | 0 | 0
  Serotype 19A | 55.6 [52.6 to 58.5] | 65.0 [62.0 to 67.8] |  |
  Serotype 22F: number analyzed (Participants) | 1099 | 1076 | 0 | 0
  Serotype 22F | 76.8 [74.2 to 79.3] | 78.5 [76.0 to 81.0] |  |
  Serotype 33F: number analyzed (Participants) | 1097 | 1067 | 0 | 0
  Serotype 33F | 71.6 [68.8 to 74.2] | 66.7 [63.8 to 69.6] |  |
  Serotype 9N: number analyzed (Participants) | 1098 | 1074 | 0 | 0
  Serotype 9N | 77.9 [75.3 to 80.3] | 29.4 [26.7 to 32.2] |  |
  Serotype 15A: number analyzed (Participants) | 1087 | 1061 | 0 | 0
  Serotype 15A | 85.7 [83.5 to 87.8] | 37.7 [34.8 to 40.7] |  |
  Serotype 15C: number analyzed (Participants) | 1095 | 1071 | 0 | 0
  Serotype 15C | 81.4 [78.9 to 83.6] | 63.2 [60.2 to 66.1] |  |
  Serotype 16F: number analyzed (Participants) | 1090 | 1074 | 0 | 0
  Serotype 16F | 81.4 [78.9 to 83.6] | 11.8 [10.0 to 13.9] |  |
  Serotype 17F: number analyzed (Participants) | 1098 | 1076 | 0 | 0
  Serotype 17F | 84.5 [82.2 to 86.6] | 4.3 [3.1 to 5.7] |  |
  Serotype 20A: number analyzed (Participants) | 1097 | 1077 | 0 | 0
  Serotype 20A | 74.7 [72.1 to 77.3] | 1.3 [0.7 to 2.2] |  |
  Serotype 23A: number analyzed (Participants) | 1091 | 1074 | 0 | 0
  Serotype 23A | 85.5 [83.3 to 87.6] | 29.4 [26.7 to 32.2] |  |
  Serotype 23B: number analyzed (Participants) | 1094 | 1075 | 0 | 0
  Serotype 23B | 76.1 [73.4 to 78.6] | 42.2 [39.3 to 45.2] |  |
  Serotype 24F: number analyzed (Participants) | 1093 | 1077 | 0 | 0
  Serotype 24F | 84.0 [81.7 to 86.1] | 2.3 [1.5 to 3.4] |  |
  Serotype 31: number analyzed (Participants) | 1094 | 1075 | 0 | 0
  Serotype 31 | 81.1 [78.6 to 83.4] | 3.9 [2.8 to 5.2] |  |
  Serotype 35B: number analyzed (Participants) | 1090 | 1075 | 0 | 0
  Serotype 35B | 83.1 [80.8 to 85.3] | 3.3 [2.3 to 4.5] |  |

13. Secondary Outcome: Percentage of Participants With ≥4-fold Change From Baseline in OPA GMTs in Cohort 1 for the Pneumococcal Serotypes Contained in V116 and PCV20
Description: Percentage of participants with ≥4-fold rise from baseline in OPA GMTs in Cohort 1 was determined using MOPA. The within-group 95% CIs were based on the exact binomial method proposed by Clopper and Pearson. The 10 common pneumococcal serotypes in both V116 and PCV20 were as follows: 3, 6A, 7F, 8, 10A, 11A, 12F, 19A, 22F, and 33F. The 11 unique pneumococcal serotypes in V116 were as follows: 9N, 15A, 15C, 16F, 17F, 20A, 23A, 23B, 24F, 31, and 35B. Per protocol, Cohort 2 were not analyzed in this outcome measure.
Time Frame: Baseline and Day 30 post-vaccination
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1 V116 | Cohort 1 PCV20 | Cohort 2 V116 | Cohort 2 PCV20
Number analyzed (Participants) | 1179 | 1177 | 0 | 0
Percentage of participants
  Serotype 3: number analyzed (Participants) | 966 | 937 | 0 | 0
  Serotype 3 | 71.3 [68.4 to 74.2] | 59.1 [55.9 to 62.3] |  |
  Serotype 6A: number analyzed (Participants) | 954 | 931 | 0 | 0
  Serotype 6A | 76.8 [74.0 to 79.5] | 79.9 [77.2 to 82.4] |  |
  Serotype 7F: number analyzed (Participants) | 967 | 961 | 0 | 0
  Serotype 7F | 71.0 [68.1 to 73.9] | 65.9 [62.8 to 68.9] |  |
  Serotype 8: number analyzed (Participants) | 999 | 971 | 0 | 0
  Serotype 8 | 75.8 [73.0 to 78.4] | 67.4 [64.3 to 70.3] |  |
  Serotype 10A: number analyzed (Participants) | 1021 | 978 | 0 | 0
  Serotype 10A | 71.9 [69.0 to 74.6] | 74.1 [71.3 to 76.9] |  |
  Serotype11A: number analyzed (Participants) | 890 | 889 | 0 | 0
  Serotype11A | 70.0 [66.9 to 73.0] | 61.5 [58.2 to 64.7] |  |
  Serotype 12F: number analyzed (Participants) | 1031 | 1022 | 0 | 0
  Serotype 12F | 89.0 [87.0 to 90.9] | 87.1 [84.9 to 89.1] |  |
  Serotype 19A: number analyzed (Participants) | 1024 | 990 | 0 | 0
  Serotype 19A | 64.4 [61.3 to 67.3] | 70.2 [67.2 to 73.0] |  |
  Serotype 22F: number analyzed (Participants) | 936 | 935 | 0 | 0
  Serotype 22F | 70.5 [67.5 to 73.4] | 74.4 [71.5 to 77.2] |  |
  Serotype 33F: number analyzed (Participants) | 937 | 938 | 0 | 0
  Serotype 33F | 67.7 [64.6 to 70.7] | 61.5 [58.3 to 64.6] |  |
  Serotype 9N: number analyzed (Participants) | 920 | 978 | 0 | 0
  Serotype 9N | 64.7 [61.5 to 67.8] | 19.9 [17.5 to 22.6] |  |
  Serotype 15A: number analyzed (Participants) | 693 | 706 | 0 | 0
  Serotype 15A | 66.7 [63.0 to 70.2] | 35.8 [32.3 to 39.5] |  |
  Serotype 15C: number analyzed (Participants) | 952 | 937 | 0 | 0
  Serotype 15C | 83.4 [80.9 to 85.7] | 74.2 [71.2 to 76.9] |  |
  Serotype 16F: number analyzed (Participants) | 910 | 961 | 0 | 0
  Serotype 16F | 71.9 [68.8 to 74.8] | 20.8 [18.3 to 23.5] |  |
  Serotype 17F: number analyzed (Participants) | 862 | 952 | 0 | 0
  Serotype 17F | 75.8 [72.7 to 78.6] | 9.5 [7.7 to 11.5] |  |
  Serotype 20A: number analyzed (Participants) | 1003 | 1011 | 0 | 0
  Serotype 20A | 67.3 [64.3 to 70.2] | 9.6 [7.8 to 11.6] |  |
  Serotype 23A: number analyzed (Participants) | 758 | 734 | 0 | 0
  Serotype 23A | 78.9 [75.8 to 81.7] | 36.8 [33.3 to 40.4] |  |
  Serotype 23B: number analyzed (Participants) | 1021 | 1021 | 0 | 0
  Serotype 23B | 85.5 [83.2 to 87.6] | 49.6 [46.4 to 52.7] |  |
  Serotype 24F: number analyzed (Participants) | 925 | 872 | 0 | 0
  Serotype 24F | 80.5 [77.8 to 83.0] | 6.3 [4.8 to 8.1] |  |
  Serotype 31: number analyzed (Participants) | 912 | 954 | 0 | 0
  Serotype 31 | 76.5 [73.6 to 79.3] | 17.9 [15.5 to 20.5] |  |
  Serotype 35B: number analyzed (Participants) | 917 | 988 | 0 | 0
  Serotype 35B | 60.0 [56.7 to 63.2] | 6.8 [5.3 to 8.5] |  |

ADVERSE EVENTS:
Time Frame: All-cause mortality (ACM): Randomization up to 194 days post-vaccination. Serous adverse events (SAEs): Treatment (Day 1) up to 194 days post-vaccination. Non-serious AEs (NSAEs): Treatment (Day 1) up to 30 days post-vaccination.
Description: ACM population for Cohorts 1 and 2 arms consisted of planned randomized participants, ACM population for the Unplanned Participants consisted of participants randomized to both V116 and PCV20. The SAE and NSAE population for Cohorts 1 and 2 aconsisted of APaT. The SAE and NSAE population for the Unplanned Participants arm consisted of participants excluded from the APaT. Participants with ACM or AEs in from the Unplanned arm were reported as zero due to the risk of identification..
Groups:
- Cohort 1: V116: Pneumococcal vaccine-naïve adult participants (≥50 years of age) receive a single dose of V116 on Day 1.
- Cohort 1: PCV20: Pneumococcal vaccine-naïve adult participants (≥50 years of age) receive a single dose of PCV20 on Day 1.
- Cohort 2: V116: Pneumococcal vaccine-naïve adult participants (18 to 49 years of age) receive a single dose of V116 on Day 1.
- Cohort 2: PCV20: Pneumococcal vaccine-naïve adult participants (18 to 49 years of age) receive a single dose of PCV20 on Day 1.
- Unplanned Participants: Participants with unplanned randomization and unplanned treatment with both V116 and PCV20.
Arm/Group | Cohort 1: V116 | Cohort 1: PCV20 | Cohort 2: V116 | Cohort 2: PCV20 | Unplanned Participants
All-Cause Mortality (participants affected / at risk) | 4/1179 | 2/1179 | 0/201 | 0/100 | 0/2
Serious Adverse Events (participants affected / at risk) | 19/1177 | 24/1175 | 1/200 | 3/100 | 0/2
Other Adverse Events (participants affected / at risk) | 615/1177 | 722/1175 | 161/200 | 78/100 | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: V116 (N=1177) | Cohort 1: PCV20 (N=1175) | Cohort 2: V116 (N=200) | Cohort 2: PCV20 (N=100) | Unplanned Participants (N=2)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery embolism (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jejunal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral mucosa erosion (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic necrosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subcapsular hepatic haematoma (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal wall abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalitis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Brain contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Radial nerve palsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device occlusion (Product Issues) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alcoholism (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Delirium tremens (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: V116 (N=1177) | Cohort 1: PCV20 (N=1175) | Cohort 2: V116 (N=200) | Cohort 2: PCV20 (N=100) | Unplanned Participants (N=2)
Fatigue (General disorders) | 240 (243) | 235 (237) | 81 (81) | 34 (34) | 0 (0)
Injection site erythema (General disorders) | 82 (83) | 86 (87) | 32 (32) | 13 (13) | 0 (0)
Injection site pain (General disorders) | 471 (474) | 608 (615) | 143 (143) | 74 (74) | 0 (0)
Injection site swelling (General disorders) | 79 (79) | 103 (105) | 28 (28) | 14 (14) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 75 (75) | 82 (83) | 33 (33) | 14 (14) | 0 (0)
Headache (Nervous system disorders) | 162 (176) | 174 (184) | 59 (62) | 26 (29) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-16): https://cdn.clinicaltrials.gov/large-docs/32/NCT05425732/Prot_SAP_000.pdf